CLINICAL TRIAL: NCT02164604
Title: Intravitreal Ranibizumab to Treat Retinopathy of Prematurity Stage 3 Plus Disease
Brief Title: Lucentis to Treat Retinopathy of Prematurity (ROP) 3 Plus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Marcel Menke, PD Dr. med univ. Marcel N Menke, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSA22-05-2014
Record Dates: First submitted 2014-05-22; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Retinopathy of Prematurity
Keywords: ranibizumab; intravitreal therapy; ROP; Plus disease; stage 3 plus
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): All eyes receive one intravitreal injection with 0.03ml ranibizumab
  Interventions: Drug: intravitreal injection of 0.03ml ranibizumab

INTERVENTIONS:
Drug: intravitreal injection of 0.03ml ranibizumab

SUMMARY:
Retinopathy of prematurity (ROP) is a neovascular retinal disorder of premature born children, characterized by the development of retinal neovascularisation, macular dragging and eventually retinal detachment. ROP is a leading cause for childhood blindness, especially in developing countries. Vascular endothelial growth factor (VEGF) plays an important role in the development of the disease. Recently, the BEAT ROP study tested the efficacy of intravitreal bevacizumab for stage 3 plus ROP in a prospective, controlled, randomized, stratified, multicenter trial. Authors found that bevacizumab showed a significant benefit for Zone I but not Zone II disease, with continuation of peripheral retinal vessel growths after treatment. The authors also concluded that safety could not be assessed due to the small sample size. Other authors raised concerns regarding the results of the BEAT ROP study and the safety of bevacizumab.

The investigators suspected a better safety profile for ranibizumab to treat stage 3 plus ROP. Here we present the outcome of 6 eyes with ROP stage 3 plus treated with a single injection of ranibizumab.

DETAILED DESCRIPTION:
The outcome of six eyes with ROP stage 3 plus treated with one single intravitreal injection of ranibizumab is presented. Safety issues and side affects are discussed. Follow up was 6 months.

ELIGIBILITY:
Inclusion Criteria:

* ROP stage 3 plus disease

Exclusion Criteria:

* Severe systemic co-morbidity that did not allow systemic sedation for injection, or were antiVEGF (vascual endothelial growth factor) therapy was contra-indicated

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
number of eyes with ocular side effects due to intravitreal ranibizumab | 6 months
  assessment of direct ocular adverse events due to intravitreal ranibizumab injections as a measure of safety

SECONDARY OUTCOMES:
number of patients with systemic side effects of intravitreal ranibizumab | 6 months
  number of patients with systemic side effects as a measure of safety.
efficacy of intravitreal ranibizumab to treat ROP stage 3 plus | 6 months
  Assessment of the regression of ROP-related changes due to treatment as a measure for efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Menke MN, Framme C, Nelle M, Berger MR, Sturm V, Wolf S. Intravitreal ranibizumab monotherapy to treat retinopathy of prematurity zone II, stage 3 with plus disease. BMC Ophthalmol. 2015 Mar 8;15:20. doi: 10.1186/s12886-015-0001-7. PMID 25886603